CLINICAL TRIAL: NCT04685226
Title: A Multicenter, Nonrandomized, Open-Label Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of ICP-723 in Patients With Solid Tumors
Brief Title: A Phase I/II Clinical Trial of ICP-723 in the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00501
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICP-723 (Experimental): ICP-723
  Interventions: Drug: ICP-723

INTERVENTIONS:
Drug: ICP-723 — ICP-723 is a white, round, uncoated table

SUMMARY:
A Multicenter, Nonrandomized, Open-Label Phase I/IIClinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of ICP-723 in Patients with Solid Tumors

DETAILED DESCRIPTION:
Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed surgically unresectable locally advanced or metastatic solid tumors or primary central nervous system (CNS) tumors..
2. Age:

   Adult Cohort: Age ≥ 18 years; Adolescent cohort: 12 ≤ years < 18 years.
3. At least one measurable lesion as per RECIST1.1 criteria, or for primary CNS tumors, at least one measurable lesion as per RANO or INRC criteria.
4. Adult cohort: ECOG PS score of 0-1;
5. Adolescent cohort: Karnofsky (age ≥ 16 years) or Lansky (age < 16 years) PS score > 60.
6. Life expectancy > 3 months.
7. Female patients or male patients of childbearing potential, who agree to use medically acceptable effective methods of birth control throughout the study up to 12 weeks after the last dose of the study treatment.
8. Patients who have signed the Informed Consent Form voluntarily and agree to follow the therapeutic regimen and the visit schedule.

Exclusion Criteria:

1. Any other active malignancy within 5 years prior to the first dose of the study drug.
2. Prior anti-cancer treatment within 28 days prior to the first dose.
3. Major surgical procedures within 4 weeks or minor surgical procedures within 2 weeks prior to the first dose of the study drug.
4. A history of allergic disease, severe drug allergy, known hypersensitivity to any component of the ICP-723 tablet formulation.
5. Other situations that, in the investigator's opinion, would make the subject unsuitable for participation in the study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2020-09-27 (Actual); Primary Completion 2028-01-25 (Estimated); Study Completion 2028-02-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 12 months
  To evaluate the safety and tolerability of ICP-723 at different doses in the treatment of advanced solid tumors;
MTD | Up to 2 Months
  To determine maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Cmax | Up to 1 month
  To preliminarily obtain pharmacokinetic (PK) data of ICP-723 in the treatment of advanced solid tumors include the peak plasma concentration (Cmax)
ORR | Up to 2 months
  Objective Response Rate

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - The First Medical Center of the Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Affiliated to Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangdong, Guangzhou
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer hospital, Changsha, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The first affiliated hospital Zhejiang university school of medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No